CLINICAL TRIAL: NCT05849233
Title: Investigating Autism Clinical Risk Factors With Profiling the Intestinal Microbiome and Metabolome Analysis and Their Impact on Disease Severity and Clinical Outcomes in Autistic Egyptian Children
Brief Title: Autism Clinical Risk Factors Investigation With Microbiome and Metabolome Profiling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: October University for Modern Sciences and Arts (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: RSPL 1.6
Record Dates: First submitted 2023-04-14; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism clinical risk factors; autism; microbiome; metabolome
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool Sample collection and storage
  * DNA Extraction
  * DNA amplification and amplicon sequencing
  * Bioinformatics processing of amplicon data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The role of gut microbiome was recently raised in the pathogenesis of neurodevelopmental disorders including autism spectrum disorder (ASD). In view of these evidences, together with poor conductance of researches on gut microbiota in ASD patients in Egypt, in addition to the absence of definite medical test or biological marker for diagnosis of ASD, the present study is designed to study clinical risk factor of autism and the predominant gut microbiome in autistic children in an attempt to identify gut bacteria which are likely related to ASD and to correlate these bacteria and clinical variables with the severity of autism. Interestingly, the totality of the studies focusing on the fecal metabolome features in ASD has investigated the differences between subjects with and without this disorder, while ignoring potential correlations between microbiome, metabolome and ASD severity

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a group of neurodevelopmental disorders characterized by impairment in communication and social interaction, and repetitive behaviors. 1%-1.5% of children in developed nations has ASD, This rate is said to range between 0.15% and 0.8% in low- and middle-income countries. Over the past decades, the prevalence of ASD has increased worldwide. Scientists have been trying to explore the molecular mechanisms behind the pathology of ASD. Several evidence suggests that genetic factors such as chromosomal abnormalities and environmental factors like diet and stress are involved in the pathogenesis and advancement of ASD. Accumulating research has demonstrated the gut-brain axis or multiple biochemical signaling pathways that take place between the gastrointestinal tract (GI tract) and the central nervous system (CNS), and its possible association with ASD. Mounting evidence explains that gut microbial dysbiosis is implicated in the pathogenesis of multiple diseases, including inflammatory bowel disease (IBS), coeliac disease (CD), and ASD. A Recent Egyptian study showed that an evidence of changes in the gut microbiome of ASD children compared to the unrelated controls. However, the microbiome profile of siblings was more like that of autistic children than that of unrelated controls. These observations may highlight the importance of the interplay between environmental and host genetic factors in shaping the gut microbiome. The study also emphasized the importance of identification of microbiome and specific microorganisms' changes that can be targeted for diagnosis as well as for treatment of ASD. This study aims to investigate clinical risk factors of autism and to elucidate the changes in gut microbiome in Egyptian autistic children and their possible correlation with clinical outcomes and the severity of the disease.

ELIGIBILITY:
Inclusion criteria:

a) Autistic children aged between 3-9 years based on DSM V

Exclusion criteria:

1. Past or present history of seizures or any other neurological illness
2. Past or present history of any psychiatric illness Those patient will be excluded to avoid confounders because those diseases also affected by microbiome The inclusion and exclusion criteria will be determined by the medical history taken from the parents of the children before test application.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Autistic children aged between 3-9 years based on DSM V with variable degrees of disease severity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Autism clinical risk factors | 1 year
  prenatal, Natal and postnatal history then regression analysis

SECONDARY OUTCOMES:
Intestinal microbiome | 1 year
  Stool Sample collection then intestinal microbiome investigation
metabolome Analysis | 1 year
  fecal metabolome analysis

CONTACTS AND LOCATIONS:
Overall Officials: sara Eladawy, PhD, Principal Investigator — MSa university; amira Abdeldaim, PhD, Study Director — MSA university
Locations (1):
- Ain shams University Hospitals (Unit of Phoniatrics-Otorhinolaryngology department ), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ahmed SA, Elhefnawy AM, Azouz HG, Roshdy YS, Ashry MH, Ibrahim AE, Meheissen MA. Study of the gut Microbiome Profile in Children with Autism Spectrum Disorder: a Single Tertiary Hospital Experience. J Mol Neurosci. 2020 Jun;70(6):887-896. doi: 10.1007/s12031-020-01500-3. Epub 2020 Feb 15. PMID 32062762